CLINICAL TRIAL: NCT06620042
Title: Functional Magnetic Resonance Imaging of Patients Receiving Intravenous Ketamine for Treatment Resistant Bipolar Depression
Brief Title: FMRI of Patients Receiving IV Ketamine for Treatment Resistant Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brian Barnett (Other)
Responsible Party: Sponsor-Investigator, Brian Barnett, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-1345
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Depression; Treatment Resistant Bipolar Depression
Keywords: ketamine; bipolar depression; bipolar disorder; bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This is a prospective open-label observational study of patients with treatment resistant bipolar depression referred for intravenous ketamine, with an interventional component of fMRI. All participants will receive an acute series of ketamine consisting of twice weekly infusions over three weeks. Non-responders will have their End of Study visits within 5 days of the last ketamine infusion. Responders (participants who achieve a ≥ 50% decrease on their QIDS-SR-16 score from Baseline) will return for three weeks of continuation treatment (weekly ketamine) and then have their End of Study visit within 5 days of the last continuation treatment. All participants will undergo fMRI prior to their first ketamine infusion and after completion of their acute series.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label Ketamine TRBD (Other): Outpatients with treatment resistant bipolar depression referred by their clinical providers for intravenous ketamine treatment
  Interventions: Drug: Ketamine; Other: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Drug: Ketamine — Open-label Ketamine
Other: Functional magnetic resonance imaging (fMRI) — Functional magnetic resonance imaging (fMRI) of the brain

SUMMARY:
This is a prospective open-label observational study of patients with treatment resistant bipolar depression referred for intravenous ketamine, with an interventional component of fMRI.

DETAILED DESCRIPTION:
This is a prospective open-label observational study of patients with treatment resistant bipolar depression referred for intravenous ketamine. All participants will receive an acute series of ketamine consisting of twice weekly infusions over three weeks. Non-responders will have their End of Study visits within 5 days of the last ketamine infusion. Responders (participants who achieve a greater than or equal to 50% decrease on their QIDS-SR-16 score from Baseline) will return for three weeks of continuation treatment (weekly ketamine) and then have their End of Study visit within 5 days of the last continuation treatment. All participants will undergo fMRI the prior to their first ketamine infusion, and after completion of their acute series.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any study related procedures are performed
2. Males/females at least 18 years of age but no older than 75 years of age
3. Meet DSM-5 criteria for a current Major Depressive Episode and lifetime Bipolar I disorder or Bipolar II disorder as determined by both:

   A. a clinician's diagnostic evaluation and B. confirmed with the MINI International Neuropsychiatric Interview (MINI 7.0.2)
4. A current depressive episode that has lasted a minimum of 4 weeks as determined by both:

   A. a clinician's diagnostic evaluation and B. confirmed with the MINI International Neuropsychiatric Interview (MINI 7.0.2)
5. Meet all the following criteria on symptom rating scales at screening:

   A. Montgomery Asberg Depression Rating Scale (MADRS) score ≥20 B. Young Mania Rating Scale (YMRS) score of ≤ 5 C. QIDS-SR-16 score of ≥ 11
6. Have had ≥ 2 adequate trials of mood stabilizers, antipsychotics (only those FDA approved for bipolar depression), or antidepressants or augmentation strategies during their lifetime. An adequate trial is defined as 4 weeks of medication at the minimum FDA approved dose.
7. In the opinion of the investigator, the patient is willing and able to comply with scheduled visits, treatment plan, and other trial procedures for the duration of the study.

Exclusion Criteria:

1. Meet DSM-5 criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, mental retardation, or pervasive developmental disorder
2. Meets any exclusion criteria for ketamine treatment (uncontrolled arterial hypertension, uncontrolled hyperthyroidism, severe ischemic heart disease or heart failure, severe liver or kidney disease, space occupying lesion in the brain or the spinal cord, and uncontrolled glaucoma)
3. The patient is pregnant or breast feeding
4. The patient has a severe medical illness or severe neurological disorder
5. The patient has a known ketamine allergy or is taking a medication that may significantly interact with ketamine (see Appendix)
6. Diagnosis of psychotic features during the current depressive episode or within the past 6 months
7. Was previously enrolled in the trial
8. Active moderate or severe substance use disorder within the last 3 months (no exclusion for tobacco use disorder of any severity)
9. Current episode of mania/hypomania or mixed episode according to MINI or study clinician
10. MRI contraindications

    * Severe head trauma
    * Claustrophobia incompatible with scanning
    * Cardiac pacemaker
    * Implanted cardiac defibrillator
    * Aneurysm brain clip
    * Inner ear implant
    * Prior history as a metal worker and/or certain metallic objects in the body -- must complete MRI screening form and be approved by MRI technologist before each scan
    * History of clinically significant vertigo middle ear disorder, or double vision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Acute Response Changes in Subgenual Cingulate Functional Connectivity | Three weeks after treatment initiation
  Seed-to-whole brain functional connectivity z-maps will be calculated from the left and right subgenual cingulate on the baseline and post-acute resting-state functional MRI (rs-fMRI) from each participant. After acute treatment, participants will be categorized as "responders" (≥50% decrease from baseline score of Quick Inventory of Depressive Symptomatology 16-item self-report, QIDS-SR-16) or "non-responders". Brain regions in responders that exhibit significantly different treatment-related change in functional connectivity compared to non-responders will be identified using general linear model methods.

SECONDARY OUTCOMES:
Acute Response Baseline Structural Connectivity | Three weeks after treatment initiation
  Baseline structural connectivity will be assessed from baseline diffusion tensor imaging for each participant. White matter tracts in responders that exhibit significantly different mean transverse diffusivity compared to non-responders will be identified.
Sustained Response Changes in Subgenual Cingulate Functional Connectivity | Six weeks after treatment initiation
  Acute "responders" will undergo a maintenance treatment phase (3 treatments over 3 weeks). After maintenance treatment, participants will be categorized as "sustained responders" (≥50% decrease from baseline QIDS-SR-16 score) or "relapsers" at the end of treatment. Brain regions in sustained responders that exhibit significantly different treatment-related change in subgenual cingulate brain functional connectivity maps compared to relapsers will be identified using general linear model methods.
Suicidal Ideation Changes in Subgenual Cingulate Functional Connectivity | Six weeks after treatment initiation
  Brain regions in participants that experience suicidal ideation during treatment that exhibit significantly different treatment-related change in subgenual cingulate brain functional connectivity maps compared to participants who do not experience suicidal ideation will be identified using general linear model methods.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Barnett, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Lutheran Hospital, Cleveland, Ohio
  - Cleveland Clinic Lutheran Hospital, Ohio City, Ohio

IPD SHARING:
Plan to Share IPD: No